CLINICAL TRIAL: NCT00678821
Title: Response and Adaptation to Aerobic Exercise in Patients With Pulmonary Hypertension: Initial Studies for Establishing Guidelines
Brief Title: Aerobic Exercise in Patients With Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: George Mason University (Other); Inova Fairfax Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 080133; 08-CC-0133
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12-03

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Pulmonary Rehabilitation
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Patients with PH will be randomized to either aerobic exercise training plus education (AET) or education only (Ed-only) treatments
  Interventions: Other: Aerobic exercise
- 2 (Active Comparator): A comparison group of patients with ILD who do not have secondary PH (ILD-only) will also undergo the AET arm
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Supervised aerobic exercise and educational lectures for 10 weeks

SUMMARY:
This study will determine if a rehabilitation exercise program can help people with pulmonary hypertension (PH) increase their physical activity. Patients with PH have an increase in blood pressure in the pulmonary blood vessels (artery, vein or capillaries) that leads to shortness of breath, dizziness, fainting and other symptoms.

Healthy volunteers and people with pulmonary hypertension between 21 and 75 years of age may be eligible for this study.

All participants undergo the following tests and procedures:

* Medical history and physical examination
* 6-minute walk test: Subjects walk as fast as they can for 6 minutes on a walking track to determine their ability to participate in physical activity.
* Questionnaires: Subjects complete nine questionnaires related to their fatigue, daily physical activity, mood, and so forth.
* Maximum treadmill test: The exercise begins at an easy level and gradually increases until the subject says he or she can no longer continue or the investigator decides it is not safe to continue. Subjects are fitted with a mask, electrodes and light sensors to measure how well the heart is working and how well the muscles use oxygen.

Patients with pulmonary hypertension undergo the following additional procedures:

* Activity monitoring: Patients wear a monitor for 3 days that measures movement and heart rate.
* Group assignment: Patients are randomly assigned to Group 1 (education plus aerobic exercise) or Group 2 (education followed by exercise).
* Group 1 patients will attend classes three days a week at either Inova Fairfax Hospital Pulmonary Rehabilitation Center or The National Institutes of Health for 10 weeks. Two sessions a week will include a 1 hour education session as well as a 30-45 minute track or treadmill exercise session. The third session will only include exercise. During the education patients will learn about a healthy lifestyle with pulmonary hypertension. After the 10 weeks of education and exercise, subjects repeat the 6-minute walk test, maximum treadmill test and questionnaires.
* Group 2 patients participate in 2; 1-hour educational session at either the Inova Pulmonary Rehabilitation Center or The National Institutes of Health for 10 weeks. After the classes, they repeat the 6-minute walk test, maximum treadmill test and questionnaires. The following 10 weeks will consist of 3 days a week of 30-45 minute track or treadmill walking at either Inova or NIH, after which they again repeat the questionnaires, treadmill and walk tests.

DETAILED DESCRIPTION:
We propose a randomized trial to determine the safety and effectiveness of aerobic exercise for patients who have primary pulmonary hypertension (PH) or PH secondary to interstitial lung disease (ILD). This project will be the first in a series of studies aimed at establishing exercise prescription and general rehabilitation guidelines for patients who have advanced lung diseases.

An essential treatment for almost all cardiovascular and pulmonary disorders is aerobic exercise training. The effectiveness of exercise rehabilitation has been established and exercise rehabilitation has become a standard of care for patients with chronic obstructive pulmonary disease (COPD). However, fundamental information about the mechanisms underlying exercise training and its therapeutic benefits remains lacking for patients who have advanced lung disease in general and specifically for those with PH.

Subjects will be over the age of 21 years. The patients will be enrolled from sites within a reasonable travel distance from the greater Washington area and will receive their exercise training at Inova Fairfax Hospital or at the National Institutes of Health (NIH) main campus. Exercise-based rehabilitation is already common for patients who have PH at the Inova Fairfax Hospital. Their pulmonary rehabilitation program is well established, and their staff is experienced in providing exercise therapy for patients with PH and advanced lung diseases. The Rehabilitation Medicine Department (RMD) at The NIH Clinical Center has established a pulmonary rehabilitation program for this protocol as well as to provide rehabilitation services for NIH clinic patients.

There will be two primary treatment arms. Patients with PH will be randomized to either aerobic exercise training plus education (AET) or education only (Ed-only) treatments. A comparison group of patients with ILD who do not have secondary PH (ILD-only) will also undergo the AET arm. Exercise training will consist of a 10-week regimen of supervised treadmill or over ground walking three times a week. Exercise session duration will be 30 minutes and will progress to 45 minutes per session over the 10 weeks. The intensity of the exercise will be between 70 and 80% of the heart rate reserve.

There will also be two secondary studies. First, the subjects with PH initially randomized to the education only arm will complete an aerobic exercise training program after participation in education. In addition, we will also compare baseline tests among patients with PH, patients with ILD-only and healthy controls.

The study outcome measures will be assessed at NIH, RMD. These will include pre- and post-exercise training comparisons of symptom limited treadmill exercise tests to assess heart rate, pulse oximetry, EKG, maximum oxygen consumption, bioelectrical impedance cardiography, and near infrared spectroscopy measurements of muscle oxygenation. We will also assess accelerometry based activity, 6-minute walk distance, and a number of other quality of life and functional measures questionnaires including: International Physical Activity Questionnaire, Fatigue Severity Scale, SF-36v2 Health Survey, Human Activity Profile, Stages of Exercise Change, Exercise Self-Efficacy, Profile of Mood States, Cambridge Pulmonary Hypertension Outcome Review.

This study represents a unique opportunity to assess the effects of exercise on patients with advanced lung disease and may open up valuable new treatment options for these patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

PH and ILD-only Groups: Subjects of this study will include individuals with ILD and PH who are referred for Pulmonary Rehabilitation. Patients with ILD, PH or PH comorbid with ILD will be included. The following list provides more specific inclusion criteria:

* Between age 21-82 years
* WHO functional class II or III, will accept WHO functional class I and IV based on 6 minute walk test results (less than or equal to 400 meters for Class I and greater than or equal to 50 meters for Class IV)
* No recent syncope or significant chest pain
* No prior Pulmonary Rehabilitation received within the last 6 months.
* Physically inactive, no participation in a structured exercise program 3 or more days a week for over 30 minutes at each session including pulmonary rehabilitation maintenance within the last 6 months.
* Patients may qualify if they have any one of the following conditions:

  * PAH diagnosed by right heart catheterization defined as resting pulmonary mean arterial pressure equal to or higher than 25 mmHg
  * Interstitial lung disease, including idiopathic pulmonary fibrosis (IPF), non-specific pulmonary fibrosis (NSPF), sarcoidosis or other form of chronic lung fibrosis will be based on clinical context via clinic note from primary pulmonologist and an echo within one year of enrollment showing an RVSP <40mmHg.

    1. If RVSP is lower than 40mmHg patients with interstitial lung disease will be enrolled without the need for a right heart catheterization.
    2. If RVSP is indeterminate on an echo procedure performed within a year of enrollment, the patient will undergo another echo test at The National Institutes of Health, Echocardiogram Laboratory.
    3. Only if RVSP is unable to be estimated on an echo at NIH, the absence of the following abnormalities on echo will be used: right ventricular enlargement, right ventricular hypertrophy, paradoxical movement of interventricular septum and/or altered pulmonary flow velocity. If RVSP is unable to be estimated and these abnormalities are absent on echo, the patient will be enrolled as an ILD-only patient. If any of these echocardiographic abnormalities are present the patient will not be enrolled until the results of a right heart catheterization can be obtained to verify the absence of pulmonary hypertension.

Healthy Controls: The controls will include individuals who have never been diagnosed with primary or secondary PH and are apparently healthy. Controls will be matched to the PH cohort for age, gender, and body mass.

* Between 21 82 years
* Physically inactive, no participation in a structured exercise program 3 or more days a week for over 30 minutes at each session.
* No cardiorespiratory or pulmonary disease
* No other diseases of the neurological, metabolic, renal, or musculoskeletal system
* No medications that would influence aerobic capacity or treadmill performance

EXCLUSION CRITERIA FOR PATIENTS WITH PH, ILD-ONLY AND HEALTHY CONTROLS:

Since the goal is to examine exercise responses and adaptations as affected by PH, patients will have no other (except the primary disease in those with secondary PH) medical conditions that would impair aerobic capacity or the ability to engage in physical activity. These conditions would include any of those affecting the cardiovascular, pulmonary, metabolic, neurological, or musculoskeletal systems. Specific exclusion criteria for the PH and control cohorts are:

* Significant Restrictive or Obstructive Lung Disease with a FEV1/FVC ratio less than or equal to 65 percent
* Diagnosis of ischemic heart disease
* Left ventricular dysfunction with the ejection fraction less than 40 or a documented pulmonary capillary wedge pressure greater than or equal to 18 mmHg.
* Acute cor pulmonale
* Dilated or hypertrophic cardiomyopathy
* Non-idiopathic cardiomyopathy
* Significant hepatic or renal dysfunction
* Metastatic cancer with a life expectance of less than 6 months
* Disabling stroke
* Active substance abuse
* Severe psychiatric disease
* Patients on Antiretroviral Therapy
* Uncontrolled diabetes mellitus with a history of DKA
* Mitochondrial disease
* Pregnancy
* Ongoing tobacco use
* Children: Individuals younger than 21 years will not be included in the protocol because reference ranges for normative aerobic capacity and aerobic fitness have not been established for these age ranges.

Ages: 21 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-06-12 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
Pre and post exercise training CPET | 10 wks
  CPET variables
Accelerometry-based activity | 10 wks
  Physical activity participation
6 minute walk distance | 10 wks
  total meters walked in 6 minutes
Quality of life and functional measures | 10 wks
  self-report questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keyser RE, Christensen EJ, Chin LM, Woolstenhulme JG, Drinkard B, Quinn A, Connors G, Weir NA, Nathan SD, Chan LE. Changes in fatigability following intense aerobic exercise training in patients with interstitial lung disease. Respir Med. 2015 Apr;109(4):517-25. doi: 10.1016/j.rmed.2015.01.021. Epub 2015 Feb 7. PMID 25698651
- [Background] Chan L, Chin LMK, Kennedy M, Woolstenhulme JG, Nathan SD, Weinstein AA, Connors G, Weir NA, Drinkard B, Lamberti J, Keyser RE. Benefits of intensive treadmill exercise training on cardiorespiratory function and quality of life in patients with pulmonary hypertension. Chest. 2013 Feb 1;143(2):333-343. doi: 10.1378/chest.12-0993. PMID 22922554
- [Background] Weinstein AA, Chin LM, Keyser RE, Kennedy M, Nathan SD, Woolstenhulme JG, Connors G, Chan L. Effect of aerobic exercise training on fatigue and physical activity in patients with pulmonary arterial hypertension. Respir Med. 2013 May;107(5):778-84. doi: 10.1016/j.rmed.2013.02.006. Epub 2013 Mar 7. PMID 23478192
- [Derived] Woolstenhulme JG, Guccione AA, Herrick JE, Collins JP, Nathan SD, Chan L, Keyser RE. Left Ventricular Function Before and After Aerobic Exercise Training in Women With Pulmonary Arterial Hypertension. J Cardiopulm Rehabil Prev. 2019 Mar;39(2):118-126. doi: 10.1097/HCR.0000000000000397. PMID 30624371
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-CC-0133.html